CLINICAL TRIAL: NCT00014586
Title: Randomized Phase III Step-Up Study On Initial Antiandrogen Monotherapy In Comparison With Watchful Waiting In Asymptomatic T1-3 Any G (Any Gleason) NO or Nx M0 Prostate Cancer Patients Without Local Treatment With Curative Intent
Brief Title: Bicalutamide Compared With Observation Followed by Bicalutamide Plus Either Goserelin or Orchiectomy in Treating Patients With Prostate Cancer
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: low accrual
Sponsor: European Organisation for Research and Treatment of Cancer - EORTC (Network)
Responsible Party: Sponsor
Allocation: Randomized | Purpose: Treatment
Other Study IDs: EORTC-30991; EORTC-GU-30991
Record Dates: First submitted 2001-04-10; First posted 2003-01-27 (Estimated); Last update posted 2012-09-24 (Estimated); Status verified 2012-09

CONDITIONS: Prostate Cancer
Keywords: stage I prostate cancer; stage IIB prostate cancer; stage IIA prostate cancer; stage III prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — bicalutamide; Goserelin; Orchiectomy

INTERVENTIONS:
Drug: bicalutamide
Drug: goserelin acetate
Procedure: orchiectomy

SUMMARY:
RATIONALE: Testosterone can stimulate the growth of cancer cells. Bicalutamide and goserelin may fight prostate cancer by reducing the production of testosterone. It is not yet known which hormone therapy regimen is most effective for prostate cancer.

PURPOSE: Randomized phase III trial to compare the effectiveness of bicalutamide with that of observation followed by bicalutamide plus either goserelin or orchiectomy for patients who have prostate cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Compare the overall and cancer-specific survival of patients with prostate cancer treated with bicalutamide alone followed by bicalutamide with either goserelin or bilateral orchiectomy vs observation followed by bicalutamide with either goserelin or bilateral orchiectomy.
* Compare the time to first and second clinical progression in patients treated with these regimens.
* Compare the quality of life, including potency, of patients treated with these regimens.

OUTLINE: This is a randomized, multicenter study. Patients are stratified according to participating center, tumor differentiation grade (G3 or Gleason more than 6 vs other values), T category, comorbidity (i.e., chronic disease) (yes vs no), potency (yes vs no), type of chosen hormonal ablation (goserelin vs orchiectomy), PSA level (less than 10 ng/mL vs 10-20 ng/mL vs 20-100 ng/mL), and N status (N0 vs NX). Patients are randomized to one of two treatment arms.

* Arm I: Patients receive oral bicalutamide once daily. At first symptomatic disease progression, patients also receive goserelin subcutaneously once every 28 or 84 days or undergo bilateral orchiectomy. At second disease progression, patients discontinue bicalutamide.
* Arm II: Patients are observed until first symptomatic disease progression. At first disease progression, patients receive bicalutamide with either goserelin or bilateral orchiectomy as in arm I. Patients discontinue bicalutamide as in arm I.

Quality of life is assessed at baseline, every 6 months for 6 years, at each disease progression, and then annually thereafter.

Patients are followed annually.

PROJECTED ACCRUAL: Approximately 1266 patients (633 per treatment arm) will be accrued for this study within 5 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed prostate cancer

  * T1-3, any G (any Gleason), N0 or NX
* High risk defined as G3 or Gleason more than 6 or PSA more than 20 ng/mL and unfit or unwilling to undergo local curative therapy OR
* Low risk defined as G1-2 or Gleason less than 7 and PSA no more than 20 ng/mL and no prior local curative therapy
* Asymptomatic (pain score of 0)
* PSA no more than 100 ng/mL (no more than 25 times normal)
* No metastatic disease by chest x-ray, bone scan (if PSA more than 10 ng/mL or 2.5 times normal), and pelvic CT (if chance of lymph node metastases is at least 5% by Partin tables)
* No bone disease that would interfere with diagnosis of metastatic disease

PATIENT CHARACTERISTICS:

Age:

* 80 and under

Performance status:

* WHO 0-2

Life expectancy:

* Not specified

Hematopoietic:

* Not specified

Hepatic:

* Not specified

Renal:

* Not specified

Other:

* No other malignancy within the past 5 years except adequately treated basal cell skin cancer
* No psychological, personal, sociological, or geographical condition that would preclude study

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Not specified

Chemotherapy

* Not specified

Endocrine therapy

* Not specified

Radiotherapy

* Not specified

Surgery

* Not specified

Max Age: 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2001-01; Primary Completion 2003-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gerald H.J. Mickisch, MD, Study Chair — Center of Operative Urology Bremen
Locations (1):
- Center of Operative Urology Bremen, Bremen, Germany